CLINICAL TRIAL: NCT00052936
Title: Randomised Study Comparing 6 And 8 Cycles Of Chemotherapy With CHOP ( Cyclophosphamide, Doxorubicin, Vincristine And Prednisone) At 14-Day Intervals (CHOP-14), Both With Or Without The Monoclonal Anti-CD20 Antibody Rituximab In Patients Aged 61 To 80 Years With Aggressive Non-Hodgkin's Lymphoma
Brief Title: Combination Chemotherapy With or Without Rituximab in Treating Older Patients With Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: German High-Grade Non-Hodgkin's Lymphoma Study Group (Other)
Responsible Party: Sponsor
Organization: Universität des Saarlandes (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000269015; DSHNHL-1999-1A (Other Grant/Funding Number: Deutsche Krebshilfe); EU-20243 (Other: Ethikkommission der Ärztekammer des Saarlandes [85/99])
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Lymphoma
Keywords: anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; stage III grade 1 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III grade 2 follicular lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage I adult lymphoblastic lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage I adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; stage I mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; contiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult Burkitt lymphoma; stage I adult Burkitt lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; contiguous stage II marginal zone lymphoma; noncontiguous stage II marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; stage I marginal zone lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, Follicular; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Burkitt Lymphoma; Lymphoma, B-Cell, Marginal Zone | interventions — Filgrastim; Rituximab; VAP-cyclo protocol; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- S6 (Experimental): 6x CHOP-14
  Interventions: Biological: filgrastim; Drug: CHOP regimen; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisone; Drug: vincristine sulfate; Radiation: radiation therapy
- R6 (Experimental): 6x CHOP-14 + 8x Rituximab
  Interventions: Biological: filgrastim; Biological: rituximab; Drug: CHOP regimen; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisone; Drug: vincristine sulfate; Radiation: radiation therapy
- S8 (Experimental): 8x CHOP-14
  Interventions: Biological: filgrastim; Drug: CHOP regimen; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisone; Drug: vincristine sulfate; Radiation: radiation therapy
- R8 (Experimental): 8x CHOP-14 + 8x Rituximab
  Interventions: Biological: filgrastim; Biological: rituximab; Drug: CHOP regimen; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisone; Drug: vincristine sulfate; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim
Biological: rituximab
  Arms: R6; R8
Drug: CHOP regimen
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: prednisone
Drug: vincristine sulfate
Radiation: radiation therapy — 36Gy on BULK and extranodal involvement

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies such as rituximab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. It is not yet known whether combination chemotherapy is more effective with or without rituximab in treating aggressive non-Hodgkin's lymphoma.

PURPOSE: This randomized phase III trial is studying how well giving cyclophosphamide, doxorubicin, vincristine, and prednisone together with or without rituximab works in treating older patients who have aggressive non-Hodgkin's lymphoma. (This trial is no longer randomized as of 6/2005).

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) with vs without rituximab in elderly patients with aggressive non-Hodgkin's lymphoma.
* Compare the efficacy of 6 vs 8 courses of CHOP chemotherapy in patients treated with these regimens.
* Compare the rate of complete remission, rate of primary progression, tumor control, disease-free survival, overall survival, and relapse after radiotherapy in patients treated with these regimens.
* Compare the safety and side effects of these regimens in these patients.

Secondary

* Compare short-term and long-term side effects of these regimens in these patients.
* Compare quality of life of patients treated with these regimens.
* Compare the cost of these regimens in these patients.
* Determine relapse in patients treated with these regimens who received involved-field radiotherapy.

OUTLINE: This is a randomized (randomized part of study completed as of 6/2005), open-label, multicenter study. Patients are stratified according to participating center, value for serum lactic dehydrogenase (no greater than upper limit of normal [ULN] vs greater than ULN), bulky disease present (no vs yes), stage (I or II vs III or IV), general ECOG status of patient (0 or 1 vs 2), and age (61 to 70 vs 71-80). Patients are randomized to 1 of 4 treatment arms. Patients with CD20-negative lymphoma are randomized to arms I or II only.

* Prephase treatment:Patients receive vincristine IV on day -6 and prednisone on day -6 to day 0 before initiating CHOP chemotherapy.
* Arm I (closed to accrual as of 7/25/2005): Patients receive standard CHOP chemotherapy comprising cyclophosphamide IV, doxorubicin IV, and vincristine IV on day 1 and oral prednisone on days 1-5. Patients also receive filgrastim (G-CSF) subcutaneously once daily on days 6-12 of each CHOP course. Treatment repeats every 2 weeks for 6 courses.
* Arm II (closed to accrual as of 7/25/2005): Patients receive standard CHOP chemotherapy and G-CSF as in arm I for a total of 8 courses.
* Arm III: Patients receive standard CHOP chemotherapy and G-CSF as in arm I. Patients also receive rituximab IV before CHOP every 2 weeks for a total of 8 courses.
* Arm IV (closed to accrual as of 7/25/2005): Patients receive standard CHOP chemotherapy and G-CSF as in arm II. Patients also receive rituximab IV before CHOP every 2 weeks for a total of 8 courses.

In all arms, treatment continues in the absence of disease progression or unacceptable toxicity.

Beginning 3-6 weeks after completion of the last chemotherapy course, after complete recovery of bone marrow, and after complete remision of mucositis, patients with sites of initial bulky disease or extranodal involvement undergo radiotherapy 5 times a week for 4 weeks.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 1580 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed aggressive non-Hodgkin's lymphoma (NHL) by an excisional biopsy of a lymph node or an extensive biopsy of an extranodal involvement (if there is no lymph node involvement)
* CD20^+ B-cell lymphoma or CD20^- B-cell and T-cell lymphoma allowed
* B-cell NHL including the following:

  * Stage III follicular lymphoma
  * Stage III follicular lymphoma and diffuse B-cell lymphoma
  * Lymphoblastic precursor B-cell lymphoma
  * Diffuse large cell B-cell lymphoma

    * Centroblastic
    * Immunoblastic
    * Plasmablastic
    * Anaplastic large cell
    * T-cell-rich B-cell lymphoma
    * Primary effusion lymphoma
    * Intravasal B-cell lymphoma
    * Primary mediastinal B-cell lymphoma
  * Mantle zone lymphoma, blastoid
  * Burkitt's lymphoma
  * Burkitt-like lymphoma
  * Aggressive marginal zone lymphoma (monocytoid)
* T-cell NHL including the following:

  * Lymphoblastic precursor T-cell lymphoma
  * Peripheral T-cell lymphoma (PTCL) not otherwise specified (NOS)

    * Lennert's lymphoma
    * T-zone lymphoma
  * T-cell lymphoma of the angioimmunoblastic lymphadenopathy with dysproteinemia (AILD) type
  * Anaplastic large cell lymphoma

    * ALK^+
    * ALK^-
  * Extranodal NK/T-cell lymphoma, nasal type
  * Intestinal T/NK-cell lymphoma (with or without enteropathy)

    * Hepatosplenic gamma-delta lymphoma
    * Subcutaneous panniculitis-like PTCL
    * Aggressive T/NK PTCL
  * Anaplastic large-cell NHL, NOS
* Bone marrow involvement no more than 25%
* No lymphoma that is clearly restricted to the CNS or originating from the gastrointestinal tract

PATIENT CHARACTERISTICS:

Age

* 61 to 80

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* WBC at least 2,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* No active hepatitis infection

Renal

* Creatinine no greater than 2 times ULN

Cardiovascular

* No Canadian Cardiovascular Society class III or IV angina pectoris
* No New York Heart Association class III or IV cardiac failure
* Ejection fraction at least 50%
* Fractional shortenings at least 25% by echocardiography or nuclear medicine examination

Pulmonary

* FEV1 at least 50%
* Diffusion capacity at least 50%

Other

* No uncontrolled diabetes mellitus
* No known hypersensitivity to any study medications
* No other concurrent malignancy
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy

Surgery

* Not specified

Other

* Must not have already initiated lymphoma therapy (except for the prephase treatment specified for this study)
* No other concurrent lymphoma therapy
* No concurrent participation in another treatment study

Ages: 61 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1506 (Actual)
Dates: Start 2001-01; Primary Completion 2010-08-05 (Actual); Study Completion 2010-08-05 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure at 3 years within the study and then periodically after study completion | 3 years within the study and then periodically after study completion

SECONDARY OUTCOMES:
Complete response rate at 3 years within the study and then periodically after study completion | 3 years within the study and then periodically after
Progression rate | 3 years within the study and then periodically after
Survival | 3 years within the study and then periodically after
Tumor control | 3 years within the study and then periodically after
Disease-free survival | 3 years within the study and then periodically after

CONTACTS AND LOCATIONS:
Overall Officials: Michael G.M. Pfreundschuh, MD, Study Chair — Universitaetsklinikum des Saarlandes
Locations (174):
- Germany (172):
  - Haematologisch Onkologische Praxis, Aachen
  - Klinikum St. Marien, Amberg
  - Gemeinschaftspraxis Fuer Innere Medizin, Haematologie Und Internistische Onkologie, Ansbach
  - II. Medizinische Klinik, Aschaffenburg
  - Specialist Practice for Oncology, Aschaffenburg
  - Haematologische Praxis, Augsburg
  - Hamatologische/Onkologische Gemeinschaftspraxis - Augsburg, Augsburg
  - Klinikum Augsburg, Augsburg
  - Kreiskrankenhaus Aurich, Aurich
  - Regional Hospital Bad Hersfeld, Bad Hersfeld
  - Humaine - Clinic, Bad Saarow
  - Krankenhaus Hohe Warte Mediziniche Klinik, Bayreuth
  - Robert Roessle Comprehensive Cancer Center - Charite Campus Buch, Berlin
  - Haematologisch-Onkologische Schwerpunktpraxis, Berlin
  - Hospital Complex Bernburg, Bernburg
  - Krankenhaus Bietigheim, Bietigheim
  - Saint Agnes Hospital, Bocholt
  - Saint Josef Hospital, Bochum
  - Knappschaft Krankenhaus, Bochum
  - Medizinische Poliklinik, Bonn
  - Rheinische Friedrich-Wilhelms-Universitat, Bonn
  - DIAKO Ev. Diakonie Krankenhaus gGmbH, Bremen
  - Medizinische Klinik Am Lukas - Krankenhaus, Bünde
  - General Hospital, Celle
  - Hospital Kuchwald Chemnitz, Chemnitz
  - Praxis Fuer Haematologie Internistische Onkologie, Cologne
  - Medizinische Universitaetsklinik I at the University of Cologne, Cologne
  - Cologne-Kalk
  - Lung Clinic Cologne-Merheim, Cologne-Merheim
  - Carl - Thiem - Klinkum Cottbus, Cottbus
  - Klinikum Darmstadt, Darmstadt
  - Saint Johannes Hospital Dortmund, Dortmund
  - Universitatsklinikum Carl Gustav Carus, Dresden
  - St. Johannes Hospital - Medical Klinik II, Duisburg
  - Franz Hospital Dulmen, Dülmen
  - Florence-Nightingale-Krankenhause, Deaconess Kaiserswerth, Düsseldorf
  - Hans - Susemihl - Krankenhaus, Emden
  - Klinikum Erfurt, Erfurt
  - St. Antonius Hospital, Eschweiler
  - Universitaetsklinikum Essen, Essen
  - Krankenhaus Nordwest, Frankfurt
  - Klinikum Frankfurt (Oder) GmbH, Frankfurt (Oder)
  - Evang. Deaconess Hospital Freiburg, Freiburg im Breisgau
  - Municipal Hospital Complex, Fulda
  - Robert - Koch Hospital, Gehrden
  - Centre for Internal Medicine Gieben, Giessen
  - Universitaetsklinikum Goettingen, Göttingen
  - Klinik Fuer Innere Medizin, Hematology/Oncology, Ernst Moritz Armdt Universitaet, Greifswald
  - Staedtisches Klinikum Guetersloh, Gütersloh
  - Allgemeines Krankenhaus Hagen, Hagen
  - St. Marien Hospital - Katholisches Krankenhaus Hagen gGmbH, Hagen
  - Krankenhaus St. Elisabeth und St. Barbara, Halle
  - Krankenhaus Martha-Maria Halle-Doelau gGmbH, Halle
  - Universitaetsklinikum Halle, Halle
  - Hamburg
  - University Medical Center Hamburg - Eppendorf, Hamburg
  - Asklepios Klinik Nord Heidberg, Hamburg
  - Allgemeines Krankenhaus Altona, Hamburg
  - Haematologisch-Onkologische Praxis Altona, Hamburg
  - Evangelische Krankenhaus Hamm, Hamm
  - Hanover
  - Henriettenstiftung Krankenhaus, Hanover
  - Krankenhaus Siloah - Medizinische Klinik II, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Oncology Specialists Clinic, Harrislee
  - Thoraxklinik Heidelberg, Heidelberg
  - Medizinische Universitaetsklinik und Poliklinik, Heidelberg
  - Regional Hospital Heidenheim, Heidenheim
  - Regional Hospital Am Plattenwald - Bad Friedrichshall, Heilbronn
  - Klinikum Herford, Herford
  - Marienhospital at Ruhr University Bochum, Herne
  - Privatklinik Dr. R. Schindlbeck GmbH & Co. KG, Herrsching am Ammersee
  - Onkologische Schwerpunktpraxis, Hildesheim
  - Evang. Hospital, Holzminden
  - Medical University Hospital Homburg, Homburg
  - Hospital Complex Hoyerswerda, Hoyerswerda
  - Gemeinschaftspraxis Innere Medizin, Jena
  - Klinikum der Friedrich-Schiller Universitaet Jena, Jena
  - Municipal Hospital Complex of the University, Kaiserslautern
  - Staedtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - Red Cross Hospital Kassel, Kassel
  - Staedtisches Krankenhaus Kiel, Kiel
  - Stiftungsklinikum Mittelrhein - Gesundheitszentrum Evangelisches Stift Sankt Martin Koblenz gGmbH, Koblenz
  - Praxis fuer Haematologie und Onkologie, Koblenz
  - Leonardis Clinic, Kornwestheim
  - Klinikum Krefeld GmbH, Krefeld
  - Frankenwald Klinik, Kronach
  - Caritas - Krakenhaus Lebach, Lebach
  - University Leipzig Clinic of Internal Medicine, Leipzig
  - Klinikum "St. Georg" Leipzig, Leipzig
  - Leipzig
  - Klinikum Lippe - Lemgo, Lemgo
  - St. Vincenz Hospital Limburg, Limburg
  - St. Bonifatius Hospital Lingen, Lingen
  - Dreifaltigkeits Hospital, Lippstadt
  - Klinikum Ludwigsburg, Ludwigsburg
  - St. Marien Hospital Ludwighafen, Ludwigshafen
  - Municipal Complex of Ludwigshafen, Ludwigshafen
  - Universitaetsklinikum Schleswig-Holstein - Campus Luebeck, Lübeck
  - Staedtisches Klinikum Magdeburg - Altstadt, Magdeburg
  - Universitaetsklinkum Magdeburg der Otto-von-Guericke-Universitaet Magdeburg, Magdeburg
  - Johannes Gutenberg University, Mainz
  - III Medizinische Klinik Mannheim, Mannheim
  - Marburg
  - Universitaetsklinikum Giessen und Marburg GmbH - Marburg, Marburg
  - Regional Hospital Mayen, Mayen
  - Klinikum Minden, Minden
  - Minden
  - Monchenglasbach/Rheydt
  - Ev. Hospital Bethesda, Mönchengladbach
  - Hospital Maria-Hilf II, Mönchengladbach
  - Munich Oncologic Practice at Elisenhof, Munich
  - Klinikum der Universitaet Muenchen - Innenstadt Campus, Munich
  - Krankenhaus Muenchen Schwabing, Munich
  - Klinikum der Universitaet Muenchen - Grosshadern Campus, Munich
  - Municipal Hospital Munich, Munich
  - Evangelisches Krankenhaus - Mulheim, Mülheim
  - St. Marien Hospital - Muelheim an der Ruhr, Mülheim
  - Kreiskrankenhaus Muenchberg, Münchberg
  - Medizinische Klinik und Poliklinik A - Universitaetsklinikum Muenster, Münster
  - Regional Hospital Neumarkt, Neumarkt
  - Staedtisches Klinikum Neunkirchen gGmbH, Neunkirchen
  - Lukaskrankenhaus Neuss, Neuss
  - Klinikum Nuernberg - Klinikum Nord, Nuremberg
  - Klinikum Offenburg, Offenburg
  - Hematologische Praxis, Oldenburg
  - Ev. Hospital Oldenburg, Oldenburg
  - Klinikum Oldenburg, Oldenburg
  - Paracelsus - Klinik Osnabrueck, Osnabrück
  - Municipal Hospital Complex, Pforzheim
  - Klinikum Ernst Von Bergmann, Potsdam
  - Kreiskrankenhaus Radebeul, Radebeul
  - Krankenhaus St. Elisabeth - Ravensburg, Ravensburg
  - Klinikum der Universitaet Regensburg, Regensburg
  - Hematologische Onkologische Praxis, Regensburg
  - Krankenhaus Barmherzige Brueder Regensburg, Regensburg
  - Jakobi Krankenhaus, Rheine
  - Klinik und Poliklinik fuer Innere Medizin - Universitaet Rostock, Rostock
  - Klinik und Poliklinik fuer Strahlentherapie - Universitaetsklinikum Rostock, Rostock
  - Rostock
  - Caritasklinik St. Theresia, Saarbrücken
  - Schwerpunktpraxis fuer Haematologie und Onkologie, Saarbrücken
  - St. Elizabeth-Klinik Saarlouis, Saarlouis
  - Martin - Luther Hospital, Schleswig
  - Deaconess Hospital, Schwäbisch Hall
  - Leopoldina - Krankenhaus, Schweinfurt
  - Evang. Jung-Stilling Hospital, Siegen
  - St. Lukas - Clinic Solingen, Solingen
  - Klinik fuer Onkologie - Katharinenhospital Stuttgart, Stuttgart
  - Diakonie Klinikum Stuttgart, Stuttgart
  - Klinikum Stuttgart - Buergerhospital, Stuttgart
  - Hospital Bad Cannstatt, Stuttgart
  - Robert-Bosch-Krankenhaus, Stuttgart
  - St. Elisabeth Hospital Thuine, Thuine
  - Regional Hospital Traunstein, Traunstein
  - Krankenanstalt Mutterhaus der Borromaerinnen, Trier
  - Trier
  - Krankenhaus Barmherzigen Brueder, Trier
  - Hospital Tutzing, Tutzing
  - Comprehensive Cancer Center Ulm at Universitaetsklinikum Ulm, Ulm
  - Ev. Hospital Unna, Unna
  - St. Marienhospital - Vechta, Vechta
  - Municipal Hospital Complex, Villingen-Schwenningen
  - Regional Hospital Waldbrol, Waldbröl
  - Evangelisches Krankenhaus Essen Werden, Werden
  - Hospital Wetzler, Wetzlar
  - Deutsche Klinik fuer Diagnostik, Wiesbaden
  - Dr. Horst-Schmidt-Kliniken, Wiesbaden
  - Ev. Hospital Witten-Herdecke, Witten
  - Kliniken St. Antonius, Wuppertal
  - University Wurzburg, Würzburg
  - Municipal Hospital Complex Zwickau, Zwickau
- Switzerland (2):
  - City Hospital Triemli, Zurich
  - UniversitaetsSpital Zuerich, Zurich

REFERENCES:
- [Result] Pfreundschuh M, Schubert J, Ziepert M, Schmits R, Mohren M, Lengfelder E, Reiser M, Nickenig C, Clemens M, Peter N, Bokemeyer C, Eimermacher H, Ho A, Hoffmann M, Mertelsmann R, Trumper L, Balleisen L, Liersch R, Metzner B, Hartmann F, Glass B, Poeschel V, Schmitz N, Ruebe C, Feller AC, Loeffler M; German High-Grade Non-Hodgkin Lymphoma Study Group (DSHNHL). Six versus eight cycles of bi-weekly CHOP-14 with or without rituximab in elderly patients with aggressive CD20+ B-cell lymphomas: a randomised controlled trial (RICOVER-60). Lancet Oncol. 2008 Feb;9(2):105-16. doi: 10.1016/S1470-2045(08)70002-0. Epub 2008 Jan 15. PMID 18226581
- [Derived] Christofyllakis K, Kaddu-Mulindwa D, Lesan V, Rixecker T, Kos IA, Held G, Regitz E, Pfreundschuh M, Bittenbring JT, Thurner L, Poeschel V, Ziepert M, Altmann B, Bewarder M. An inherited genetic variant of the CEP72 gene is associated with the development of vincristine-induced peripheral neuropathy in female patients with aggressive B-cell lymphoma. Ann Hematol. 2024 Nov;103(11):4599-4606. doi: 10.1007/s00277-024-05973-9. Epub 2024 Sep 4. PMID 39227453
- [Derived] Kuhnl A, Cunningham D, Counsell N, Hawkes EA, Qian W, Smith P, Chadwick N, Lawrie A, Mouncey P, Jack A, Pocock C, Ardeshna KM, Radford J, McMillan A, Davies J, Turner D, Kruger A, Johnson PW, Gambell J, Rosenwald A, Ott G, Horn H, Ziepert M, Pfreundschuh M, Linch D. Outcome of elderly patients with diffuse large B-cell lymphoma treated with R-CHOP: results from the UK NCRI R-CHOP14v21 trial with combined analysis of molecular characteristics with the DSHNHL RICOVER-60 trial. Ann Oncol. 2017 Jul 1;28(7):1540-1546. doi: 10.1093/annonc/mdx128. PMID 28398499
- [Derived] Pfreundschuh M, Poeschel V, Zeynalova S, Hanel M, Held G, Schmitz N, Viardot A, Dreyling MH, Hallek M, Mueller C, Wiesen MH, Witzens-Harig M, Truemper L, Keller U, Rixecker T, Zwick C, Murawski N. Optimization of rituximab for the treatment of diffuse large B-cell lymphoma (II): extended rituximab exposure time in the SMARTE-R-CHOP-14 trial of the german high-grade non-Hodgkin lymphoma study group. J Clin Oncol. 2014 Dec 20;32(36):4127-33. doi: 10.1200/JCO.2013.54.6861. Epub 2014 Nov 17. PMID 25403207
- [Derived] Bittenbring JT, Neumann F, Altmann B, Achenbach M, Reichrath J, Ziepert M, Geisel J, Regitz E, Held G, Pfreundschuh M. Vitamin D deficiency impairs rituximab-mediated cellular cytotoxicity and outcome of patients with diffuse large B-cell lymphoma treated with but not without rituximab. J Clin Oncol. 2014 Oct 10;32(29):3242-8. doi: 10.1200/JCO.2013.53.4537. Epub 2014 Aug 18. PMID 25135997
- [Derived] Held G, Murawski N, Ziepert M, Fleckenstein J, Poschel V, Zwick C, Bittenbring J, Hanel M, Wilhelm S, Schubert J, Schmitz N, Loffler M, Rube C, Pfreundschuh M. Role of radiotherapy to bulky disease in elderly patients with aggressive B-cell lymphoma. J Clin Oncol. 2014 Apr 10;32(11):1112-8. doi: 10.1200/JCO.2013.51.4505. Epub 2014 Feb 3. PMID 24493716
- [Derived] Horn H, Ziepert M, Becher C, Barth TF, Bernd HW, Feller AC, Klapper W, Hummel M, Stein H, Hansmann ML, Schmelter C, Moller P, Cogliatti S, Pfreundschuh M, Schmitz N, Trumper L, Siebert R, Loeffler M, Rosenwald A, Ott G; German High-Grade Non-Hodgkin Lymphoma Study Group. MYC status in concert with BCL2 and BCL6 expression predicts outcome in diffuse large B-cell lymphoma. Blood. 2013 Mar 21;121(12):2253-63. doi: 10.1182/blood-2012-06-435842. Epub 2013 Jan 18. PMID 23335369
- [Derived] Muller C, Murawski N, Wiesen MH, Held G, Poeschel V, Zeynalova S, Wenger M, Nickenig C, Peter N, Lengfelder E, Metzner B, Rixecker T, Zwick C, Pfreundschuh M, Reiser M. The role of sex and weight on rituximab clearance and serum elimination half-life in elderly patients with DLBCL. Blood. 2012 Apr 5;119(14):3276-84. doi: 10.1182/blood-2011-09-380949. Epub 2012 Feb 15. PMID 22337718